CLINICAL TRIAL: NCT06117683
Title: Non-inferiority Comparative Trial Between Sotair® Device Attached to Manual Resuscitator Versus Mechanical Ventilation in Patients Undergoing Non-emergent Surgery With General Anesthesia
Brief Title: Non-inferiority Trial Between Sotair® Device Attached to Manual Resuscitator Versus Mechanical Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Mark Kendall, Director of Clinical Research, Rhode Island Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1963885
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Airway Management; Respiration, Artificial
Keywords: Mechanical Ventilation; General Anesthesia; Bag Mask Ventilation; Adult Sotair Device
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Study Design A non-inferiority trial; a pre-post study design (single group, within-group comparison)
Who Masked: Care Provider
Masking Description: The care provider will not know the recorded lung function recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bag mask ventilation with Adult Sotair device (Active Comparator): The anesthesia provider will manually bag ventilate with the Adult Sotair® device for 3 minutes.
  Interventions: Device: ADULT Sotair Device
- Mechanical Ventilation (No Intervention): The anesthesia provider will remove the bag valve mask and Adult Sotair® device and connect the patient to the mechanical ventilator. The recording of pressure and flow will last for 3 minutes.

INTERVENTIONS:
Device: ADULT Sotair Device — Sotair® device employs a flow limiting and pressure control valve mechanism.
  Other Names: Sotair; SafeBVM
  Arms: Bag mask ventilation with Adult Sotair device

SUMMARY:
Effective respiratory ventilation is achieved by moving the right amount of air in and out of the lungs while keeping the pressures at a safe level. A disposable safety device, Adult Sotair®, was created to improve manual ventilation delivery. In this non-inferiority study, we will perform a pre-post study design (single group, within-group comparison) to test the non-inferiority of the Adult Sotair® device compared to mechanical ventilation.

DETAILED DESCRIPTION:
Poor manual ventilation technique is a well-documented problem which occurs irrespective of a provider's qualifications or experience. A disposable safety device, Adult Sotair®, was created to improve manual ventilation delivery among providers. The device is attached to a bag valve mask (i.e. manual resuscitator) and employs a flow limiting valve mechanism to minimize excessive pressure in the airway system without venting air by capping peak flow rates at 55 L/min. For an average adult with normal lung compliance and resistance, this corresponds to a maximum airway pressure of approximately 20 cmH2O which minimizes air entry into the stomach. In this non-inferiority study, a pre-post study design (single group, within-group comparison) to test the non-inferiority of the Adult Sotair® device compared to mechanical ventilation with respect to airway pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are scheduled for non-emergency surgery with general anesthesia at Rhode Island Hospital.
* American Society of Anesthesiologists physical status 1 and 2

Exclusion Criteria:

* ASA PS >3 (e.g., respiratory disease)
* Oropharyngeal or facial pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Peak airway pressure | Recorded for 3 minute duration for each arm of the study
  mean peak airway pressure expressed in cm H20

SECONDARY OUTCOMES:
Tidal volume | Recorded for 3 minute duration for each arm of the study
  The amount of air that moves in or out of the lungs with each respiratory cycle. Measured in mL.
Airflow | Recorded for 3 minute duration for each arm of the study
  Represents the volume of air moved per unit of time during inspiration and expiration. Measured s
Respiratory rate | Recorded for 3 minute duration for each arm of the study
  The number of breaths. Measured as breaths per minute.
Oxygen saturation (SpO2) | Recorded for 3 minute duration for each arm of the study
  A present of oxygen-bound hemoglobin in the blood.
End Tidal CO2 | Recorded for 3 minute duration for each arm of the study
  The level of carbon dioxide at the end of an exhaled breath. Expressed as a percentage of CO2 or mmHg.
Blood pressure | Recorded for 3 minute duration for each arm of the study
  Is the measurement of the pressure or force of blood inside your arteries. Measured as mm Hg.
Heart rate | Recorded for 3 minute duration for each arm of the study
  The number of times your heart beats per minute. Measured as beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kendall, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD that underlie results in a publication will be shared with other researchers.
Supporting Information: SAP
Time Frame: The SAP will be available at the end of the trial for three years. The data that supports the findings of this study will be available from the corresponding investigator upon reasonable request.

REFERENCES:
- [Background] Fogarty M, Kuck K, Orr J, Sakata D. A comparison of controlled ventilation with a noninvasive ventilator versus traditional mask ventilation. J Clin Monit Comput. 2020 Aug;34(4):771-777. doi: 10.1007/s10877-019-00365-1. Epub 2019 Jul 23. PMID 31338661
- [Background] von Goedecke A, Bowden K, Wenzel V, Keller C, Gabrielli A. Effects of decreasing inspiratory times during simulated bag-valve-mask ventilation. Resuscitation. 2005 Mar;64(3):321-5. doi: 10.1016/j.resuscitation.2004.09.003. PMID 15733761
- [Background] Culbreth RE, Gardenhire DS. Manual bag valve mask ventilation performance among respiratory therapists. Heart Lung. 2021 May-Jun;50(3):471-475. doi: 10.1016/j.hrtlng.2020.10.012. Epub 2020 Nov 1. PMID 33138977
- [Background] Hutten MC, Goos TG, Ophelders D, Nikiforou M, Kuypers E, Willems M, Niemarkt HJ, Dankelman J, Andriessen P, Mohns T, Reiss IK, Kramer BW. Fully automated predictive intelligent control of oxygenation (PRICO) in resuscitation and ventilation of preterm lambs. Pediatr Res. 2015 Dec;78(6):657-63. doi: 10.1038/pr.2015.158. Epub 2015 Aug 31. PMID 26322409
- See also: Adult Sotair Products — https://safebvm.com